CLINICAL TRIAL: NCT06338410
Title: Impact of Kangaroo Mother Care on Selected Bio Marker and Maternal-Infant Bonding in Preterm Neonates in a Tertiary Care Hospital of Lahore, Pakistan
Brief Title: Effect of Kangaroo Mother Care on Oxidative Stress and Bonding
Acronym: KMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Collaborators: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Samreen Manzoor, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHS/Education/126-24/131
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Kangaroo Mother Care; Oxidative Stress
Keywords: Bonding; Kangaroo mother care; Oxidative Stress; Prematurety; Allantoin
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KMC group (Experimental): Premature infants and their mothers who will be provided with kangaroo mother care on third day of life. baby will be placed on bare chest of mother and before and after KMC urine samples will be collected from premature infants.
  Interventions: Behavioral: Kangaroo Mother Care
- Control group (No Intervention): premature infants and their mothers who will be provided with same conventional incubator care in NICU on day third of life their urine samples will also be collected before and after conventional care

INTERVENTIONS:
Behavioral: Kangaroo Mother Care — KMC is a care system for LBW and preterm infants at birth, based on skin-to-skin contact between the infant and the mother and exclusive breast feeding. The mother carries her Preterm infant for at least one hour per day. Urine collected before and after skin-to-skin contact.
  Arms: KMC group

SUMMARY:
The goal of this clinical trial is to learn if Kangaroo Mother care can have effect on oxidative stress in premature neonates. It will also learn about the bonding between mother and her premature infant. The main questions it aims to answer are:

* Does Kangaroo mother care lower the biomarker of oxidative stress in premature neonates?
* Is Kangaroo mother care associated with mother-infant bonding? Researchers will compare Kangaroo mother care to Conventional incubator care to see if Kangaroo mother care works to have effect on oxidative stress.

Participants will be:

* given Kangaroo mother care on third day of life or standard incubator care for one hour
* Urine sample for oxidative stress biomarker will be collected via noninvasive method before and after Kangaroo mother care or conventional incubator care from premature neonates.
* Mother-infant bonding scale will be filled by mothers of enrolled premature infants before and after kangaroo mother care and conventional incubator care

DETAILED DESCRIPTION:
Researcher will follow existing guidelines for shifting of infant from incubator to the mother's chest. The researcher will assist the mothers to have the baby from the incubator and to sit in the special KMC chair and bed. Urine will be collected from premature infants before and after KMC/Incubator care on third day of life by applying urine collection bag. This method is highly successful in collecting urine non-invasively. Collected urine is then placed in ice box till transportation to lab at University of Health sciences(UHS). and stored at -80 °C. After completion of data collection enzyme-linked immunosorbent assay ELISA kit of Oxidative stress biomarker (Allantoin) will be used for checking level of Allantoin in stored samples within a week. Mothers of both the KMC and control groups will be given the Mother-infant bonding scale (MIBS) self-rating instrument on 3rd Day postpartum before and after KMC and incubator care for bonding assessment.

ELIGIBILITY:
Inclusion Criteria:

* For Pre-term Neonates:

  1. 24-36 weeks' gestation Premature infants
  2. Medically stable as determined by a Score of Neonatal Acute Physiology & Perinatal Extension (SNAPPE-II); pre-term neonates with score of less than 9.
  3. Both gender
  4. Weight 1.5kg to 2.499 kg

For Mothers of Pre-term Neonates:

1. Medically stable Mothers.

Exclusion criteria:

The criteria for exclusion will be as follows:

For Pre-term Neonates:

Those will be excluded who are with below given conditions:

1. Require any kind of surgery.
2. Intraventricular hemorrhage (IVH) > or equal to grade 3.
3. On medication such as morphine, fentanyl, midazolam, muscle relaxants, phenobarbital.
4. Severe cyanotic heart disease or severe RDS.
5. Abdominal wall or intestinal anomaly or injury.
6. Chromosomal Disorder
7. Facial anomaly.

For Mothers of Pre-term Neonates:

1. Mothers having Complications of delivery like Post partem hemorrhage.
2. Any acute illness
3. Complicated cesarean section

Ages: 3 Days to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
biomarker of Oxidative Stress (Allantoin) in urine sample of premature infants | OnThird day of life before and after one hour of KMC or Conventional care
  Biomarker of oxidative stress (Allantoin) in urine samples of premature infants by ELISA Testing before and after one hour session of KMC by ELIZA testing
Mother- Infant Bonding | OnThird day of life before and after one hour of KMC or Conventional care
  by Using Mother Infant bonding self rating scale (MIBS) of eight points descriptors bonding between mother and her infant will be measured. Total scores range from 0 to 24. A high score indicates worst mother to infant bonding.

CONTACTS AND LOCATIONS:
Overall Officials: Samreen Manzoor, MSN, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Services Hospital, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data that will be published in research article. Data will be available to other researchers. data of all participants after analysis will be included in research article.
Time Frame: After publication data will be available and available till infinite time
Access Criteria: criteria will be uploaded after the publication of this research